CLINICAL TRIAL: NCT00468052
Title: Use of Dexmedetomidine Infusion for Analgesia and Emergence Agitation for Children Undergoing Tonsillectomy and Adenotonsillectomy
Brief Title: Decrease Emergence Agitation and Provide Pain Relief for Children Undergoing Tonsillectomy & Adenoidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0120060313
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2015-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; tonsillectomy; adenoidectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl (Active Comparator): fentanyl bolus 1ug.kg-1
  Interventions: Drug: fentanyl
- dexmedetomidine (Experimental): dexmedetomidine 2ug.kg-1 over 10 min followed by 0.7ug.kg-1.h-1
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — 2 micrograms/kilogram as a bolus then 0.7 micrograms/kilogram infusion
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: fentanyl — 1 microgram/kilogram as a bolus
  Other Names: Sublimaze
  Arms: fentanyl

SUMMARY:
Pediatric tonsillectomy (with or without adenoidectomy) is a brief but painful surgery carried out in children who very often also present with obstructive sleep apnea. To provide pain relief, i.e. analgesia, current practice relies on opioids , e.g., morphine or fentanyl. These narcotics are known to depress respiration and to increase the incidence of post-operative nausea and vomiting. These side effects are worrisome in this patient cohort. An alternative medication, dexmedetomidine, may have an opiate sparing effect and has a high safety profile in adults as well as in sedation in children. The purpose of this study is to determine if intravenous dexmedetomidine given as an infusion during general anesthesia for tonsillectomy or adenotonsillectomy reduces the incidence and severity of emergence agitation, improves analgesia and reduces nausea and vomiting in the 60 minutes following surgery.

DETAILED DESCRIPTION:
Emergence agitation (EA) from general anesthesia is a frequent phenomenon in children age 1-10 yrs recovering from anesthesia that demands increasing nursing care in the PACU, delays reunion with parents and often causes dissatisfaction for parents, and may lead to adverse sequelae in some cases such as physical harm to the child, in particular to the site of surgery (1). Emergence agitation is a state of non purposeful restlessness an inconsolability. This state is often accompanied by thrashing, screaming, prolonged crying and disorientation. Children are generally unaware of their surroundings and cannot be consoled by the caregivers/parents. It is very disturbing for parents to observe this behavior in their children. It is also a safety issue for children and staff. These negative effects of EA have motivated clinicians to investigate possible etiologies and potential treatments for EA.

EA may be in part due to the relative paucity of inhibitory neurotransmitters in children's central nervous system (CNS). As well, all modern anesthetics have been designed to be rapidly eliminated resulting in abrupt change from a state of anesthesia to a state of responsiveness. The result is a difficult problem managing these patients over a 30-50 minute period following pediatric anesthesia.

We propose studying patients scheduled for tonsillectomy or adenotonsillectomy. Adenotonsillar hypertrophy may produce upper airway obstruction, dysphagia, dental malocclusion, altered orofacial growth, altered eustachian tube function, or pulmonary hypertension with cor pulmonale. Obstructive sleep apnea (OSA) is associated with loud snoring during sleep with periods of respiratory pauses terminated with gasping and agitated arousal and has been suggested to have developmental consequences including ADHD, failure to thrive, and nocturnal enuresis (2). Obstructive sleep apnea syndrome is most commonly associated with adenotonsillar hypertrophy and more children are now presenting for adenotonsillectomy (3). Tonsillectomy and adenotonsillectomy are highly successful in eliminating OSA in children and is considered first-line therapy if the family is amenable and there are no specific contraindications, and is approximately 85-95% effective in eliminating OSA in children (4). All children undergoing tonsillectomy or adenoidectomy should be considered to be at increased risk for perioperative airway problems (5). Opioids may cause respiratory depression, and thus present an added risk in patients undergoing tonsillectomy and adenotonsillectomy, especially in children with OSA (6).

The purpose of this study is to determine if intravenous dexmedetomidine given as an infusion during general anesthesia for tonsillectomy or adenotonsillectomy reduces the incidence and severity of emergence agitation in the 60 minutes following surgery compared to normal practice. A second outcome is whether the need for intra-operative and postoperative analgesic narcotic medications is reduced.

Dexmedetomidine, a specific alpha 2-adrenergic receptor agonist, has recently been studied for its sedative, amnestic, and analgesic properties and has been shown to be effective in providing sedation, decreased anesthetic requirements during surgery and in postanesthesia care units, and reduction in emergence agitation (7, 8, 9). Dexmedetomidine has been shown to enhance the analgesic action of nitrous oxide and furthermore it has also been shown to be effective as a total intravenous anesthetic agent in certain patients if doses are increased to a high enough level, with no respiratory depression (10, 11). If dexmedetomidine can be shown to reduce or eliminate emergence agitation, and provide effective intraoperative and postoperative analgesia without respiratory depression, this would give anesthesiologists a better option in the management of patients undergoing tonsillectomy and adenotonsillectomy.

The dosing regimen for Dexmedetomidine in a loading dose of 1ug/kg with with a continuous infusion of 0.2-0.7 ug/kg is recommended for sedation in the Intensive Care Unit for adults. There is an increasing body of experience with use of Dexmedetomidine in pediatrics both for sedation and to reduce kg/hr. They observed a mean decline in heart rate (HR) and blood pressure (BP) from pre-sedation values of 15%, with 70% of patients showing a decline between 1-30%. Despite the drop in HR and BP, all changes were still within the clinical range of normal for age (10). We are proposing 2 ug/kg as a loading dose with a maintenance dose of 0.7ug/kg/hr during surgery, since we intend to use dexmedetomidine during tonsillectomy and adenotonsillectomy, a surgery which can stimulate a pain response and the surgery starts soon after the patient is intubated with no surgical preparation time . 2ug/kg is higher than the usual recommended dose, but has been used in children in the above study without any significant adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ages 2-10 ASA rating of I-III undergoing general anesthesia tonsillectomy with and without adenoidectomy

Exclusion Criteria:

* diagnosis of anxiety disorder or chronic pain syndrome chronic disabilities or developmental delays are currently on psychotherapeutic or sedating medication are on chronic pain medication or opiate any known adverse effect to the study drug any known cardiac abnormalities

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Patel, MD, Principal Investigator — University of Medicne & Dentistry of New Jersey
Locations (1):
- UMDNJ University Hospital, Newark, New Jersey, United States

REFERENCES:
- [Background] Isik B, Arslan M, Tunga AD, Kurtipek O. Dexmedetomidine decreases emergence agitation in pediatric patients after sevoflurane anesthesia without surgery. Paediatr Anaesth. 2006 Jul;16(7):748-53. doi: 10.1111/j.1460-9592.2006.01845.x. PMID 16879517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period April 2007 to June 2009.Children recruited from the practice of the same pediatric otolaryngologist at UH in Newark. The study was introduced to the parent/legal guardian during the preoperative visit. Consent was obtained on the morning of surgery by a member of the pediatric anesthesiology study team.
Pre-assignment Details: None as long as the subject fit the inclusion criteria
Groups:
- Fentanyl (F) Group: 61 subjects in group F received IV (1mcg/kg)as a bolus as soon as IV access was established.
  0
- Dexmedetomidine: 61 subjects Group D received IV dexmedetomidine 2mcg/kg over 10 minutes followed by an infusion of 0.7mcg.kg/hr
Period: Overall Study
Arm/Group | Fentanyl (F) Group | Dexmedetomidine
Started | 68 (1 subject withdrew consent.Surgery was cancelled for 2. 4 subjects eliminated for break in protocol) | 69 (One had an intraoperative complication and was withdrawn. 7 eliminated for a break in protocol.)
Target Enrollment | 70 | 70
Completed | 61 | 61
Not Completed | 7 | 8
Not completed — Protocol Violation | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl (F) Group | Dexmedetomidine | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 61 | 122
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (1.5) | 4.2 (2.1) | 4.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 35 | 35 | 70
Region of Enrollment [Number; unit: participants]
  United States | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Emergence Agitation and Pain
Description: emergence agitation and pain will be assessed. Pediatric Anesthesia Emergence Delirium Scale (PAED) range 0-20 a lower score indicates the child is calm and the higher score indicates severe agitation. Cole Agitation Scale was employed which is a 5 point Likert scale. Parameters ranging 1 to 5 1=child is calm and 5 =the child is severly agitated .
  Objective Pain Score range is 0-10 (higher score the greater pain). 3 Parameters are captured systolic b/p,crying, movements, agitation , complaints of pain
Time Frame: On arrival to PACU and 2 hours postoperatively
Population: per protocol, OPS, PAED and Cole scale are expressed as median values of the maximum score
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fentanyl (F) Group | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
units on a scale
  PAED | 14 [0 to 20] | 10 [0 to 20]
  Cole EA | 4 [1 to 5] | 3 [1 to 5]
  OPS | 5 [0 to 10] | 3 [0 to 10]
Statistical Analysis 1: Comparison: Fentanyl (F) Group vs Dexmedetomidine; Sixty subjects were required per group to determine that with Dex would decrease the incidence of severe EA after surgery by 50% with 80% power (0.05)in comparison with the control group.60 subjects were required by group to show the that intraoperative rescue fentanyl and rescue morphine in the PACU would be 50% lower in subjects receiving dex; Test type: Superiority or Other; p = .001, Wilcoxon (Mann-Whitney) — Null hypothesis is not significantly different from group D and F
Statistical Analysis 2: Comparison: Dexmedetomidine; Null hypothesis dexmedetomidine would be a safe and effective substitute to opiates in reducing pain and the incidence of severe EA; Test type: Non-Inferiority or Equivalence — Treatment with Dex would reduce the incidence of severe agitation be 50% with an 80% power (alpha 0.05); p = .001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Duration of Agitation
Description: Cole EA scale 1=calm , 5=unconsolable
Time Frame: on arrival to PACU and for 2 hours postoperatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fentanyl | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
minutes | 11.85 (12.02) | 6.59 (7.42)
Statistical Analysis 1: Comparison: Fentanyl vs Dexmedetomidine; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Hemodynamic Stability
Description: Participants whose heart rate per minute was below 60 intraoperatively. Participants whose systolic blood pressure dremonstrated < 30% decrease from baseline and sustained for 5 minutes received rescue as defined by the protocol.
Time Frame: intraoperatively
Measure: Number; unit: participants
Arm/Group | Fentanyl (F) Group | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
participants
  heart rate below 60 bpm | 0 | 0
  systolic blood pressure <30% below baseline | 0 | 0

4. Secondary Outcome: Time to Awaken
Description: defined as spontaneous eye opening or on command
Time Frame: at end of surgery
Population: per protocol
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fentanyl (F) Group | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
minutes | 8.75 (4.06) | 7.18 (4.05)
Statistical Analysis 1: Comparison: Fentanyl (F) Group vs Dexmedetomidine; Test type: Superiority or Other; p = 0.03, Fisher Exact

5. Secondary Outcome: Time to Extubation
Description: defined as time from end of surgery to tracheal extubation
Time Frame: at end of surgical procedure
Population: per protocol
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fentanyl (F) Group | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
minutes | 10.44 (4.15) | 8.59 (4.51)
Statistical Analysis 1: Comparison: Fentanyl (F) Group vs Dexmedetomidine; Test type: Superiority or Other; p = 0.02, Fisher Exact

6. Secondary Outcome: Number of Participants With SpO2 < or Equal to 95%
Time Frame: on arrival to PACU and 2 hours postoperatively
Measure: Number; unit: participants
Arm/Group | Fentanyl | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
participants | 2 | 4

7. Secondary Outcome: Participants Requiring Morphine Rescue in PACU
Time Frame: arrival in PACU to 2 hours postoperatively
Measure: Number; unit: participants
Arm/Group | Fentanyl | Dexmedetomidine
Number analyzed (Participants) | 61 | 61
participants | 25 | 11

ADVERSE EVENTS:
Time Frame: 24 hours.
Description: At the end of surgery but prior to extubation the subject demonstrated symptoms of pulmonary edema. She was treated with lasix, chest x-ray done. It was elected to keep the pt intubated overnight in an ICU unit. She was extubated the following day and did very well.
Groups:
- Fentanyl (F) Group: No subjects in group F experienced an adverse event.
  0
- Dexmedetomidine: 1 subjects Group D experienced an adverse event.
Arm/Group | Fentanyl (F) Group | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl (F) Group (N=61) | Dexmedetomidine (N=61)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — At the end of the surgical procedure and prior to extubation the pt exhibited symptoms of pulmonary edema which was confirmed by x ray. It was elected to keep the child intubated and observe for 24 hours in ICU setting. Discharge the following day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes